CLINICAL TRIAL: NCT05064995
Title: The Bipolar Disorder in the Longitudinal Course- Genom-wide Analysis of the genotype1 - phenotype2- Relationships in the Longitudinal Course of Psychosis
Brief Title: BIPLONG - The Bipolar Disorder in the Longitudinal Course
Acronym: BIPLONG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 25-355 ex 12/13
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with the Diagnosis of a Bipolar Disorder
- Healthy Controls: Individuals with no diagnosis of Bipolar Disorder

SUMMARY:
The BIPLONG (The Bipolar Disorder in the Longitudinal Course ) study is a longitudinal study on the course of bipolar disorders and comprises two sub-studies: On the one hand, BIPLONG examines the genetic foundation and change in bipolar disorder, on the other hand, metabolic changes, clinical symptoms and cognition in bipolar disorders is evaluated. A current subproject of BIPLONG is the analysis of the psychological response of the COVID-19 (Corona virus disease) pandemic. With the parameters examined in BIPLONG, it is hoped to gain better understanding of the bipolar disorder in the longitudinal course.

DETAILED DESCRIPTION:
Study Procedure:

In addition to the bipolar patients, healthy controls will also be included. The same inventories will be used for the control subjects and the same examinations or visits will be performed; bipolar-specific disease questions will not be asked in controls.

Intervention: Longitudinal study

Method:

All patients and controls undergo several assessments every six months:

Blood samples are collected with the following main parameters of interest being examined:

* Collection and analysis of DNA, establishment of permanent cell lines, determination of mRNA and gene products (proteins), proteomics, lipidomics.
* Routine parameters: Blood count, TSH, T3, T4, homocysteine, creatinine, amylase, lipase, CK, urea, uric acid, coagulation, HBA1c, glucose, lipids (triglyceryl, LDL, HDL, cholesterol, mass spectrometry), transaminases, CRP- levels, vitamin D.
* Biomarkers: oxidative stress parameters and antioxidants, neuroinflammatory markers (e.g. interleukins, tumor necrosis factor, interferons, GDNF, VEGF, etc.), neurotrophins (BDNF, NT, Trk..), insulin, IGF, adipokines, Apo-E and AAT analysis, tryptophan/kynurenine metabolites
* Intestinal hormones grehlin, glucagon-like peptides 1 and 2 (GLP-1/2) and cholecystokinin

Additionally, socio-demographic data and psychological data are collected by administering self-assessment questionnaires. Further, neurocognitive tests are administered.

The current psychological and psychiatric state of all subjects is examined by external ratings done by experts.

Anthropomethric measures are examined (waist-to-hip ratio, blood pressure, weight, height).

Additionally, MRI is conducted on all subjects (for patients every 6 months, for controls every 12 months).

Primary hypothesis:

* Gene-environment interactions are significantly contributory to bipolar affective disorder.
* There are pathologically altered neurobiological markers that play a role in the pathogenesis of bipolar disorder.
* There is an influence of anthropometric data on the course of bipolar disorder.

Statistical analysis and anticipated sample size:

Baseline data analysis will be investigated using a multi-factorial between subject design, with the variables of group (bipolar patients versus healthy controls), gender (males versus females), weight (normal weight versus overweight), etc. as independent factors, depending on the research question. As dependent variables, in addition to sociodemographic and clinical variables (number of episodes, etc.), physiological parameters (blood parameters, anthropometry and lipometer data, EEG, ECG, MRI) and psychological variables (psychological questionnaires) will be investigated. Likewise, covariates such as age or body mass index will be included as needed.

Correlation analyses (bivariate, partial) should show possible correlations between the variables. Discriminant analyses should find out which variable best separates the investigated groups (e.g. patients vs. controls). Furthermore, regression analyses (linear, multiple) will be performed to obtain additional information about the predictive value of the variables under investigation. All analyses will be computed using IBM SPSS Statistics 20.

For the "a priori analysis" of the follow-up study (T1-T5), a repeated measures design (repeated measures within factors) was adopted. The case number calculation (effect size d between .30 and .80; Cohen, 1988) for the F-test thus results in a sample size of 47 patients with a target effect size of .40 (power 95%; alpha .05; calculated with GPower 3.1). The correlation analyses at the first measurement time point (power .95, alpha .05, effect size: .35) yields 79 subjects per group (Pat. vs. controls) at all time-points.

ELIGIBILITY:
Inclusion criteria:

* Pat. with bipolar disorder, with an age between 18 and 85 years.
* Euthymic/ maximum mildly depressed at the time of consent (for this, the severity of depression will be determined using the Hamilton Depression Scale, this will also be included in any calculations).

Exclusion criteria:

* Pat. refuses participation
* Currently severely depressed/manic episode at the time of consent
* Other currently active severe mental/ brain organic disease (epilepsy, brain tumor..)
* St.p. severe craniocerebral trauma/ brain surgery.
* Reduced intelligence (IQ< 70)
* Moderate/ severe dementia (Mini Mental Status Examination, MMSE, 20 and above)
* Clearly substance-induced clinical picture

Inclusion criteria healthy controls:

* For the whole procedure, made controls (age, gender) are needed. For this purpose we recruit controls by word of mouth or ask relatives of bipolar patients if they would like to participate. Patients are tested for the presence of a possible mental illness using Mini-DIPS (Diagnostisches Interview bei psychischen Störungen)
* Inclusion criteria: 18-75 years, no severe mental illness (depression, mania, psychosis; severe anxiety or obsessive-compulsive disorder requiring treatment, addictive disorder other than nicotine).

Exclusion criteria:

* First-degree relatives with severe mental illness.
* Severe active drug dependence (i.e. alcohol, benzodiazepines morphines)
* Current major depressive/ manic episode
* Other currently active severe mental/ brain illness (epilepsy, brain tumor..)
* St.p. severe craniocerebral trauma/ brain surgery.
* Congenital/ early childhood acquired intelligence impairment
* Moderate/ severe dementia (from MMSE 20)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bipolar disorder and healthy controls within the age frame of 18-75 are included.
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2013-06-13 (Actual); Primary Completion 2022-06-13 (Estimated); Study Completion 2022-06-13 (Estimated)

PRIMARY OUTCOMES:
CVLT- california verbal learning test | at six months
  The California Verbal Learning Test (CVLT) provides a brief and individualized assessment of verbal learning strategies and processes. The higher the score, the better the outcome
STROOP Farbe-Wort-Interferenz-Test (FWIT) | at six months
  As an objective and reliable multidimensional performance test, the Color-Word. The Interference Test measures elementary information processing skills (selection, encoding, and decoding) in the visual-verbal functional domain. The lower the score, the better the outcome.
D2-R | at six months
  To measure the subject's ability to concentrate and the speed and accuracy in distinguishing similar visual stimuli. The higher the score, the better the outcome.
"Reading the eyes of the mind" =Theory of mind | at six months
  measurement of the ability to detect social cues. The higher the score, the better the outcome.
Trail Making Test A/B, TMT-A | at six months
  Measurement of cognitive processing speed, as well as linguistic, executive, and attentional components. The lower the score, the better the outcome.
Mehrfachwahl Wortschatz Test (MWT-B) | at six months
  Measurement of the general intelligence level. The higher the score, the better the outcome.
Number Symbol Test | at six months
  Measurement of processing speed. The higher the score, the better the outcome.
Number Repeat | at six months
  Measurement of working memory. The higher the score, the better the outcome.
Beck Depressions Inventar II (BDI-II) | at six months
  Measurement of depression severity; 21 items on a scale of 0-3 (ascending). The higher the score, the worse the outcome.
Manie-Selbstbeurteilungsskala (MSS) (self-rating scale) | at six months
  Measurement of manic symptoms; 48 items (dichotomous). The higher the score, the worse the outcome.
Questionnaire of religiosity | at six months
  socio-demographic assesment of religiosity; 2 items.
Big Five Inventory-10 (BFI-10) | at six months
  Measurement of personality variables; 10 items on a scale of 1-5 (ascending).
World Health Organisation Quality of Life (WHOQOL Bref) | at six months
  Measurement of life-quality and health; 26 items on a scale of 1-5 (ascending).
Life Event Questionnaire (LEQ) | at six months
  Measurement of life events and their influence; 79 items on a scale of 0-3 (ascending)
Temperament and affective disorders (TEMPS-A)-Scale | at six months
  35 items on a scale of 1-5 (ascending). The higher the score, the better the outcome.
Brief symptom inventory (BSI) | at six months
  Measurement of psychological symptoms; 53 items on a scale of 0-4 (ascending). The higher the score, the worse the outcome.
Anhedonia scale (AS) | at six months
  Measurement of Anhedonia; 14 items on a scale of 1-4 (ascending). The higher the score, the worse the outcome.
Maslach Burnout Inventory (MBI-GS-D) | at six months
  Measurement of burnout symptoms; 16 items on a scale of 1-6 (ascending). The higher the score, the worse the outcome.
Resources in Sexuality and Partnership (RSP) | at six months
  Measurement of relationship emotions; 25 items on a scale of 1-5 (ascending).The higher the score, the better the outcome.
Satisfaction in the couple relationship (ZIP) | at six months
  Measurement of relationship satisfaction; 7 items on a scale of 1-5 (ascending), 3 items open questioned. The higher the score, the better the outcome.
Demographic Data | at six months
  Measurement of demographic data
Questionnaire of current life situation | at six months
  Measurement of demographic and diagnostic data;
Anthropometric Data - weight | at six months
  Measurement of weight
Anthropometric Data- height | at six months
  Measurement of height
Anthropometric Data - waist-to-hip ratio | at six months
  Measurement of waist-to-hip ratio
Anthropometric Data - blood pressure | at six months
  Measurement of blood pressure
Clinical Global Impression (CGI) | at six months
  External rating of a symptom severity; 2 items on a scale of 0-7 (ascending). The higher the score, the better the outcome.
Global Assessment Scale of Functioning (GAF) | at six months
  External rating of level of functioning; 1 item on a scale of 1-100 (ascending). The higher the score, the better the outcome.
Hamilton Depression Scale (HAMD) | at six months
  External rating of depression symptoms; 21 items on a scale of 0-4 (ascending).The higher the score, the worse the outcome.
Young Mania Rating Scale (YMRS) | at six months
  External rating of manic symptoms; 11 items on a scale of 0-4/0-8 (ascending). The higher the score, the worse the outcome.
Specific Level of Functioning Assessment and Physical health Inventory (SLOF) | at six months
  External rating of functioning; 43 items on a scale of 1-5 (ascending), 2 items open questioned. The higher the score, the better the outcome.
Supplementary Data for External Rating | at six months
  External rating of bipolar symptoms; 7 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria